CLINICAL TRIAL: NCT01381848
Title: An Open-Label Study to Evaluate the Single-Dose Pharmacokinetics, Safety, and Tolerability of Doripenem in Infants (Term and Preterm), Less Than 12 Weeks Chronological Age
Brief Title: A Study of Doripenem in Infants Less Than 12 Weeks of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CR016192; DORIPED1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-04-21; First posted 2011-06-27 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Bacterial Infections
Keywords: Doripenem; DORIPED1003; Intravenous; Infection; Colonization; Prophylaxis; Pediatric; Antibiotic; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Doripenem Type=exact number unit=mg/kg number=5 form=solution for injection route=intravenous use once on Day 1 for patients <8 weeks CA.,Doripenem Type=exact number unit=mg/kg number=8 form=solution for injection route=intravenous use once on Day 1 for patients >=8 weeks CA.
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — Type=exact number, unit=mg/kg, number=5, form=solution for injection, route=intravenous use, once on Day 1 for patients <8 weeks CA.
Drug: Doripenem — Type=exact number, unit=mg/kg, number=8, form=solution for injection, route=intravenous use, once on Day 1 for patients >=8 weeks CA.

SUMMARY:
The purpose of this study is to measure drug levels of doripenem in blood samples collected before and after administration of doripenem to infants less than 12 weeks of age who are hospitalized and documented, presumed to have, or are at risk for bacterial infection (s) and are undergoing treatment with intravenous (i.v.) antibiotics. Safety and tolerability will also be assessed.

DETAILED DESCRIPTION:
This is a multicenter, open-label (identity of treatment is known to patient's parent/legal guardian/caregiver and to all study staff) pharmacokinetic study (a study to observe how the drug is absorbed and distributed within the body) to measure drug levels of doripenem in hospitalized but medically stable infants (term and preterm), <12 weeks of chronological age (CA) (age since time of birth) who have documented, presumed to have, or are at risk for bacterial infection(s) and are undergoing treatment with intravenous (i.v.) (administered in a vein) antibiotics. Doripenem will be administered alone at any time after the first dose of a nonstudy antibiotic is administered to the patient. Doripenem is not being used in this study to treat infection and it will not replace the patient's prescribed antibiotic(s). The duration of the study will be up to 9 days for each patient. Patients' safety will be monitored throughout the study by a safety committee who will review safety information at least once a month or after every 8 patients are enrolled and dosed. Safety evaluation will include, but will not be limited to, adverse events, clinical laboratory tests, and vital signs. A single dose of study drug (doripenem) will be administered to patients in a hospitalized setting. Patients <8 weeks CA will receive a 5 mg/kg doripenem 1-hour i.v. infusion, and patients >=8 weeks CA will receive an 8 mg/kg doripenem 1-hour infusion. Study drug will be administerd to the patient alone at any time after the first dose of a nonstudy antibiotic is administered to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Must be hospitalized, medically stable, without acute decline in physical condition in the inestigator's judgement
* Documented, presumed to have, or are at risk for bacterial infection(s) and are undergoing treatment with i.v. antibiotics
* Patient's weight (kg) must be within the 5th and the 95th percentile inclusive for his or her age
* Parent or the patient's legally acceptable representative must have signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to allow the infant to participate in the study

Exclusion Criteria:

* Clinically significant abnormal values for hematology or clinical chemistry at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination or vital signs at screening, as deemed appropriate by the investigator
* Patients who, in the investigator's judgment, have compromised renal (kidney) function including renal failure
* History of clinically significant allergies to medications, especially known hypersensitivity or intolerance to carbapenems, penicillins, or other beta lactam antibiotics
* Known allergy to heparin or history of heparin-induced thrombocytopenia, if an indwelling cannula (e.g., heparin lock) or central line is used
* Patients concomitantly treated with or having received imipenem/cilastin within 48 hours before study drug administration

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Doripenem concentrations in blood samples | Before and after study drug administration for 1 day

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to Day 7
Changes in clinical laboratory test results | From Day -2 to Day 1
Changes in vital signs measurements | From Day -2 to Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (7):
  - Little Rock, Arkansas
  - Orange, California
  - Royal Oak, Michigan
  - New Brunswick, New Jersey
  - Toledo, Ohio
  - Houston, Texas
  - Salt Lake City, Utah
- Leuven, Belgium
- United Kingdom (5):
  - Chertsey
  - Exeter
  - Liverpool
  - Manchester
  - Norwich

REFERENCES:
- [Derived] Cirillo I, Vaccaro N, Castaneda-Ruiz B, Redman R, Cossey V, Bradley JS, Allegaert K. Open-Label Study To Evaluate the Single-Dose Pharmacokinetics, Safety, and Tolerability of Doripenem in Infants Less than 12 Weeks in Chronological Age. Antimicrob Agents Chemother. 2015 Aug;59(8):4742-9. doi: 10.1128/AAC.00485-15. Epub 2015 May 26. PMID 26014957